CLINICAL TRIAL: NCT06569550
Title: Neuromodulation of the Left Premotor Cortex With Transcranial Magnetic Stimulation to Alleviate Fatigue in Multiple Sclerosis - a Randomised Controlled Clinical Trial
Brief Title: Fatigue Alleviation Through Neuromodulating Therapy in Multiple Sclerosis
Acronym: FANTiMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Research Centre for Magnetic Resonance (Other)
Collaborators: Danish Multiple Sclerosis Center (Unknown); Scleroseforeningen (Unknown); Independent Research Fund Denmark (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FANTiMS
Record Dates: First submitted 2024-08-12; First posted 2024-08-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Fatigue
Keywords: Transcranial Magnetic Stimulation, Repetitive; Magnetic Resonance Imaging; Magnetic Resonance Imaging, Spectroscopy
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Fatigue

STUDY DESIGN:
Intervention Model Description: Randomized (1:1) parallel group study to either active treatment or sham
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The TMS stimulation machine (MagPro XP orange edition, MagVenture A/S, Farum, Denmark), in combination with an A/P-coil with a separate active and placebo (sham) side. The sham side is designed to deliver <5% of the magnetic field of the active side, with similar tactile and auditory input.
  The coil is designed to be reversible, with no markings as to which side is which. There is an internal sensor that allows the device to determine which side is up. Masking is ensured by a pre-programmed code, unique to each participant, which is input in the device whereafter the device will indicate if the "wrong" side is being used for stimulation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Repetitive Transcranial Magnetic Stimulation (rTMS) (Active Comparator): Active Repetitive Transcranial Magnetic Stimulation (rTMS)
  Interventions: Device: Real Repetitive Transcranial Magnetic Stimulation
- Sham Repetitive Transcranial Magnetic Stimulation (Sham Comparator): Sham Repetitive Transcranial Magnetic Stimulation
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Real Repetitive Transcranial Magnetic Stimulation — Five sessions of real paired-pulse rTMS at 0.72Hz (inter-pulse interval of 30ms and inter-pair interval of 1381ms), for a total of 1300 pulse-pairs (30 minutes), across 5 sequential days, Monday to Friday.
  The stimulation is applied with a MagPro XP Orange stimulator (MagVenture A/S, Farum, Denmark), through a B65-Cool-A/P-CO coil (Magventure A/S) with an active and placebo (sham) side. The active side is an actively cooled figure-of-eight coil with an outer diameter of 65mm.
  Intensity is 80% of resting motor threshold. It is kept the same across all 5 sessions.
  The target is the left PMd, at MNI coordinates (34, -2, 66), transformed into patient space. Optimal coil placement, with respects to induced e-field at the target coordinates, is simulated with SimNIBS, based on the participants own MR images. The coil positioning is guided and monitored continuously with a neuronavigation system (Localite, Bonn, Germany) and the aid of robotic arm (Axilum Robotics, Schiltigheim, France ).
  Arms: Active Repetitive Transcranial Magnetic Stimulation (rTMS)
Device: Sham Repetitive Transcranial Magnetic Stimulation — Five sessions of real paired-pulse rTMS at 0.72Hz (inter-pulse interval of 30ms and inter-pair interval of 1381ms), for a total of 1300 pulse-pairs (30 minutes), across 5 sequential days, Monday to Friday.
  The stimulation is applied with a MagPro XP Orange stimulator (MagVenture A/S, Farum, Denmark), through a B65-Cool-A/P-CO coil (Magventure A/S) with an active and placebo (sham) side. The sham side does not deliver a magnetic pulse to the participant.
  The target is the left PMd, at MNI coordinates (34, -2, 66), transformed into patient space. Optimal coil placement, with respects to induced e-field at the target coordinates, is simulated with SimNIBS, based on the participants own MR images. The coil positioning is guided and monitored continuously with a neuronavigation system (Localite, Bonn, Germany) and the aid of robotic arm (Axilum Robotics, Schiltigheim, France ).
  Arms: Sham Repetitive Transcranial Magnetic Stimulation

SUMMARY:
The goal of this clinical trial is to learn if repetitive Transcranial Magnetic Stimulation (rTMS) of the left premotor cortex can lessen fatigue in patients with Multiple Sclerosis, and if this is a feasible intervention. It will also give further information on fatigue in Multiple Sclerosis. The main questions it aims to answer is:

* Does premotor rTMS decrease fatigue symptoms in patients with Multiple Sclerosis?
* Is the change in fatigue reflected in an altered balance between brain excitation and inhibition in the targeted premotor cortex?

Researchers will compare real rTMS with sham rTMS (which does not stimulate with a magnetic field), to see if real rTMS works to alleviate fatigue.

Participants will:

* Receive real or sham rTMS for 30 minutes, 5 days in a row
* Visit the clinic before and 6 days after for baseline and follow-up
* Fill out on-line questionnaires 1 day and 4 weeks after the end of intervention
* Undergo a total of 3 brain scans (Magnetic Resonance Imaging at ultra-high field), at baseline, end of intervention, and follow-up
* Undergo lab neurophysiological measurements before and after the first intervention session
* Keep a fatigue diary and wear an activity tracker in the period before and after the intervention

DETAILED DESCRIPTION:
BACKGROUND:

Multiple sclerosis (MS) is an immune mediated disease, targeting the central nervous system. Globally, the prevalence and incidence are increasing. It is a chronic condition, with no known definitive cure. Fatigue is among the most disabling MS symptoms, and is highly prevalent afflicting up to 78%-95% of patients. Fatigue in persons with MS (PwMS) is consistently associated with lower quality of life and severity of fatigue is generally associated with employment status, and may worsen over time.

PATHOPHYSIOLOGY:

The pathophysiological basis for fatigue in MS is poorly understood, with several possible contributors. However, trait fatigue in everyday life associates with task-related hyperactivation of the premotor cortex during a non-fatiguing grip force task. Patients who are able to increase premotor activity after performing a fatiguing motor task are less affected by fatigue during everyday life. Taken together, these findings support the hypothesis, that patients suffering from trait fatigue allocate their premotor "neural resources" less efficiently than patients without fatigue. This implies a mismatch in the physiological neuronal inhibition/excitation balance, and is evident as hyperactivity of the premotor cortex during "normal" motor activities, which in turn impedes an efficient upscaling of premotor activity.

CURRENT TREATMENTS:

Currently, the pharmacological treatment options for MS-related fatigue are limited and unsatisfactory. Neither of the 2 commonly used pharmaceutical agents, Amantadine nor Modafinil, show both a significant and a clinically relevant reduction in fatigue. Physical exercise has an overall positive, and clinically relevant, effect on MS-related fatigue, but physical therapy is not a feasible intervention for all PwMS. Evidence from TMS studies of the motor-cortex in fatigued PwMS, suggests that this effect may be mediated by changes in motor network excitability.

RTMS:

Repetitive Transcranial Magnetic Stimulation (rTMS) is a non-invasive method for inducing plastic focal changes in the brain. It has been investigated for multitudes of ailments, and is considered a generally safe intervention. rTMS has been repeatedly shown to have a direct and lasting neuromodulating effect on the motor cortex after stimulation of the premotor network. It is suggested that inhibitory rTMS targeting the dorsal premotor cortex can improve motor performance.

PREVIOUS TRIALS:

While rTMS is extensively investigated in other contexts, there exists few studies on MS-related fatigue. A single small study (n=33), focused on safety, targeting either motor cortex or prefrontal cortex with an H-coil, failed to show a significant effect of the intervention. Several studies have shown an effect on fatigue as a secondary outcome. However, the heterogeneity in interventional protocol and target prevents further analysis. As far as the investigators are aware, no studies have investigated alleviating fatigue by neuromodulation of the premotor network.

OBJECTIVES:

The investigators will conduct a double-blinded randomized controlled trial, investigating the effect of rTMS in fatigue in PwMS. The investigators will conduct clinical measurements for their primary outcome. Clinical outcomes will be supported by ultra-high field MRI and neurophysiological measurements, as well as supplementary clinical outcomes, in order to acquire a broad dataset for further illumination of mechanisms. For outcomes, see relevant section.

STUDY DESIGN:

The trial consists of a baseline period; an intervention period; and a follow-up period.

At the baseline visit (D0), all participants will undergo clinical testing; structural 7T MRI; 7T MR Spectroscopy (MRS) to acquire baseline neurometabolite concentrations; functional connectivity (rs-fMRI) and structural connectivity (DWI). Between D0 and the first intervention day, participants will wear a wrist-borne accelerometer and fill out a fatigue diary.

The intervention period consists of 5 sequential weekdays, Monday through Friday. On the first day of treatment (D1), neurophysiological measures of motor excitation/inhibition will be acquired before and immediately after the intervention, using single- and paired-pulse TMS, with electromyography (EMG) as a readout. On the fifth and last intervention day (D5), participants will undergo immediate follow-up 7T MRI with metabolic, functional- and structural connectivity measures.

The main follow-up is 6 days after the last rTMS session, day 11 counting from first intervention. Here they will undergo follow-up clinical testing, follow-up 7T MRI with metabolic, functional- and structural connectivity measures. Between D5 and the Follow-up, participants will again wear a wrist-borne accelerometer and fill out a fatigue diary. At first day after end of intervention, and at 4 weeks after end of intervention, participants will be invited to fill out electronic questionnaires of relevant patient-reported outcomes.

CRITERIA FOR DISCONTINUATION:

Patients are discontinued in the study in case of inability to perform a baseline MRI scan; occurrence of MS relapse; new occurrence of any condition that is a contraindication for rTMS; excessive lack of compliance to the experimental protocol as assessed by the experimenters. Additionally, all subjects reserve the right to, at any time, withdraw from the study for any reason.

QUALITY ASSURANCE:

This is a one-site study, and will be monitored by an internal monitoring process, akin to Good Clinical Practice guidelines. All procedures will be done according to a pre-defined protocol, ensuring a standard operating procedure for acquisition of all data.

Additionally. The MR- and EMG-data quality is inspected during and right after data acquisition, as is normal practice in the clinical routine and research.

Logbooks are kept for all sessions and all deviations from protocol will be noted. Data quality is further assessed through the subsequent offline data processing stage, through standardized processing pipelines.

All staff who perform MR and TMS have received comprehensive training in the respective methods, as well as safety training. All staff involved in the project will be familiar with the procedure and methods and trained the experimental procedure before conducting measurements.

DATA ANALYSIS PLAN:

Primary outcome: All patients who attend at least one rTMS session and have follow-up data available, will be included in the intention-to-treat analysis for the primary outcome, regardless of amount of rTMS sessions completed.

EMG and MRI data will be preprocessed by a blinded researcher according to standardized pipelines. For EMG data, all trials will be manually checked by a blinded researcher for muscle artefacts preceding the TMS pulse, and offending trials removed.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of relapse-remitting or secondary progressive multiple sclerosis, according to most recent McDonald's criteria (Thompson et al., 2018). This diagnosis must not be more recent than 3 months
* Must have fatigue as a complaint, and an FSMC score corresponding to at least moderate fatigue (>53)
* Stable MS medication for at least 3 months

Exclusion Criteria:

* Pregnancy, any subject with the potential to become pregnant must ensure against this (e.g. by taking oral contraceptives, or other high efficacy method)
* MS Relapse or steroid treatment within 3 months prior to inclusion
* Current treatment targeted towards fatigue, or previous if discontinued within 3 months prior to inclusion
* History of neurologic disease or other significant medical conditions, aside from MS
* EDSS > 6.5
* Major psychiatric disorder, including current clinical depression.
* Intake of medication that primarily acts on CNS or neurotransmission, except SSRI or SNRI
* Pacemaker or other implanted electronic devices
* Any intracranial metal
* Any metallic implant incompatible with MR scanning
* Claustrophobia
* Either patient or their close relatives suffering from epilepsy
* Current Drug or alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in patient reported fatigue severity, measured by the Fatigue Scale for Motor and Cognitive Symptoms (FSMC) from baseline to +6 days | Follow-up at 6 days post intervention. Compared to baseline
  Difference in change in score in Fatigue Scale for Motor and Cognitive functions, between baseline and clinical follow-up, between real and sham group.
  It is a validated 20 item score, designed for fatigue in MS. It has motor and cognitive subscales. Range 20-100. Cut-off for mild, moderate and severe fatigue is 43, 53 and 63 respectively.

SECONDARY OUTCOMES:
Change from baseline in regional brain tissue concentration of glutamate/glutamine in the stimulated premotor cortex, measured by single-voxel Magnetic Resonance Spectroscopy | Day 5 of intervention and 6 days post end of intervention, compared to baseline
  Difference in change in concentration in metabolites, measured using Ultra High Field MR Spectroscopy, between baseline and day 5 of the intervention and clinical follow-up. Between real and sham group.
  Glutamate and Glutamine are some of the major excitatory neurotransmitters. It is measured as an outcome to assess the inhibitory load in the premotor/motor system.
  At lower fields, they are often combined (to Glx) due to difficulties in separating them. At 7T this is typically not necessary.
Change from baseline in Brain tissue concentration of GABA in the stimulated premotor cortex, measured by single-voxel Magnetic Resonance Spectroscopy | Day 5 of intervention and 6 days post end of intervention, compared to baseline
  Difference in change in concentration in metabolites, measured using Ultra High Field MR Spectroscopy, between baseline and day 5 of the intervention and clinical follow-up. Between real and sham group.
  GABA is one of the major inhibitory neurotransmitters. It is measured as an outcome to assess the inhibitory load in the premotor/motor system.
Change from baseline in patient reported fatigue severity, measured by the Fatigue Scale for Motor and Cognitive Symptoms (FSMC) | Follow-up at 1 and 28 days post intervention. Compared to baseline.
  Difference in change in score in Fatigue Scale for Motor and Cognitive functions, between baseline and questionnaire follow-up, between real and sham group. Changes in fatigue score at other time points, than main follow-up, will be treated as a secondary outcome.
  It is a validated 20 item score, designed for fatigue in MS. It has motor and cognitive subscales. Range 20-100. Cut-off for mild, moderate and severe fatigue is 43, 53 and 63 respectively.
Change from baseline in objective fatiguability, measured by the Fatiguability Index (FI) | Follow-up at 6 days post intervention. Compared to baseline.
  Difference in change in fatiguability (state fatigue) measured as fatiguability index (FI). FI is calculated based on a sustained 30s maximum voluntary contraction, where FI is defined as the ratio between the actual area under the curve over the theoretical max if 100% had been sustained for the entire contraction. Range 0-1.
Change from baseline in patient-reported fatiguability, measured by the Pittsburgh Fatiguability Score (PFS) | Follow-up at 1, 6 and 28 days post intervention. Compared to baseline.
  Pittsburgh Fatiguability Score (PFS) is a self-reported rating scale of fatiguability. It contains 10 activities, each scored from 0-5 (5 being worst) for both induced cognitive and physical fatigue.
  The investigators have no specific hypothesis for the score at 1 day post intervention due to the retrospective aspect of this score.

OTHER OUTCOMES:
Change from baseline in patient reported physical fatigue severity, measured by the Fatigue Scale for Motor and Cognitive Symptoms (FSMC), physical subscore | Follow-up at 1, 6 and 28 days post intervention. Compared to baseline.
  Difference in change in score in Fatigue Scale for Motor and Cognitive functions, for the 2 physical and cognitive subscores, between baseline and questionnaire follow-up, between real and sham group. Changes in fatigue score subscores will be treated as secondary outcomes.
  It is a validated 20 item score, designed for fatigue in MS. It has 10 items each for motor and cognitive subscales. Range 10-50.
Change from baseline in patient reported cognitive fatigue severity, measured by the Fatigue Scale for Motor and Cognitive Symptoms (FSMC), cognitive subscore | Follow-up at 1, 6 and 28 days post intervention. Compared to baseline.
  Difference in change in score in Fatigue Scale for Motor and Cognitive functions, for the 2 physical and cognitive subscores, between baseline and questionnaire follow-up, between real and sham group. Changes in fatigue score subscores will be treated as secondary outcomes.
  It is a validated 20 item score, designed for fatigue in MS. It has 10 items each for motor and cognitive subscales. Range 10-50.
Per-session changes in patient reported fatigue using the Visual-Analogue Fatigue Scale (VAFS) | Time-series, 5 intervention days.
  Difference in change in fatigue, by VAFS scale, before/after each intervention, across the 5 intervention sessions. Participants will self-assess fatigue by a VAS scale before and after each intervention.
  Asking before and after at each sessions allows differentiation between acute effects due to the intervention, and effects that consolidate between sessions.
Change from baseline in patient-reported depression symptoms, measured with the Major Depression Inventory (MDI) | Follow-up at 6 days post intervention. Compared to baseline.
  MDI depression score is a commonly used rating scale for depressive symptoms. Range 0-50. Cut-offs for mild-, moderate- and severe depression are 21, 26 and 31 respectively.
Change from baseline in motor-network functional connectivity, measured by resting state functional MRI | Day 5 of intervention and 6 days post end of intervention, compared to baseline
  Resting state (rs-) Blood-oxygen level dependent (BOLD-) functional (f-) Magnetic Resonance Imaging (MRI) is a method for quantifying functional connectivity. The investigators will analyze the functional connectivity within the premotor-motor network, and how this connectivity changes as a result of the intervention.
  An exploratory framework to illuminate mechanisms of fatigue will be employed.
Change from baseline in motor network structural connectivity, measured by Diffusion Weighted Imaging | Day 5 of intervention and 6 days post end of intervention, compared to baseline.
  Diffusion Weighted Imaging (DWI) is a special MR technique to describe brain microstructure, most commonly white matter fiber direction and integrity. The investigators will analyze the structural connectivity within the premotor-motor network, and how this connectivity changes as a result of the intervention.
  An exploratory framework to illuminate mechanisms of fatigue will be employed.
Change from baseline in patient reported sleep quality, measured by the Epworth Sleepiness Scale (ESS) | Follow-up at 1, 6 and 28 days post intervention. Compared to baseline.
  Difference in change in Epworth Sleepiness Scale. The ESS is a well-validated and often used score of sleepiness, used across many different fields. The range is from 0-24 and a score above 10 usually indicated a dysfunction of sleep.
Change from baseline in patient-reported symptom severity, measured by the Multiple Sclerosis Impact Scale (MSIS-29) | Follow-up at 1, 6 and 28 days post intervention. Compared to baseline.
  Multiple Sclerosis Impact Scale (MSIS-29) is a self-reported rating scale for the impact of MS on daily quality of life. It contains 29 items, scored from 1-5 (5 being worst).
Per-session patient reported side-effects, with the TMS Adverse Events and Associated Sensations Questionnaire (TMS-SENS-Q) | Time-series, 5 intervention days.
  The TMS Adverse Events And Associated Sensations Questionnaire (TMS-SENS-Q) will be used to ask participants to self-report side-effects of rTMS after each rTMS intervention. It asks participants to self-report severity, onset and duration of 20 potential symptoms of TMS, including "other".
Change from baseline in bimanual dexterity, measured with the 9-hole peg test (9HPT) | Follow-up at 6 days post intervention. Compared to baseline.
  Cohort description, exploratory. Difference in change in scores in 9-hole peg test. The 9HPT is well-validated and often used test of fine motor function. The score consists of the average completion time across 2 trials per hand. There exists normative material, stratified by age.
Change from baseline in processing speed, measured with the Symbol Digit Modalities Test (SDMT) | Follow-up at 6 days post intervention. Compared to baseline.
  Cohort description, exploratory. Difference in change in scores in Symbol Digit Modalities Test. The SDMT is a well-validated and often used cognitive test, generally considered to assess processing speed. The score is the total number of symbols correctly assigned a number via a pre-determined key, in 90 seconds. There exists normative material, stratified by age.
Change from baseline in ambulation speed, measured with the Timed 25ft walk test (T25FW) | Follow-up at 6 days post intervention. Compared to baseline.
  Cohort description, exploratory. Difference in change in scores in 25ft walk test. The T25FW is a well-validated and often used test to assess walking ability. The score is the average time taken to walk 25ft across 2 trials. There exists normative material, stratified by age.
Change from baseline in visual memory, measured with the Brief Visual Memory Test, revised edition (BVMT-R) | Follow-up at 6 days post intervention. Compared to baseline.
  Cohort description, exploratory. Difference in change in scores in BVMT-R. The BVMT-R is a well-validated and often used test to assess short term visual memory, in MS. The score is the sum of remembered visual cues across 3 trials, in accordance with BICAMS guidelines. There exists normative material, stratified by age.
Change from baseline in verbal memory, measured with the California Verbal Learning Test (CVLT) | Follow-up at 6 days post intervention. Compared to baseline.
  Cohort description, exploratory. Difference in change in scores in CVLT. The CVLT is a well-validated and often used test to assess short term verbal memory, in MS. The outcome is the sum og words recalled across the 5 initial trials, in accordance with BICAMS guidelines. There exists normative material, stratified by age.
Multiple Sclerosis related disability, measured by the Extended Disability Status Scale (EDSS) at baseline | One-time measurement at baseline.
  Used for proper cohort description when reporting. The EDSS is a clinical rating scale ranging from 0 (no symptoms or objective signs of disability related to Multiple Sclerosis) to 10 (death caused by Multiple Sclerosis).
Change across 1 intervention session in measured Intracortical Inhibition (SICI) | Day 1, measurements done immediately (within 1 hour) before and after the intervention
  Difference in change between real and sham group, in intracortical inhibition (SICI) measured with paired-pulse TMS-EMG.
  The SICI is the ratio between the amplitude of a motor-evoked potential from 2 TMS pulses delivered at 80% and 120% of the resting motor threshold at an interval of 2.5ms, and a control potential evoked by a single pulse at 120% of resting motor threshold.
Change across 1 intervention session in measured Intracortical Facilitation (ICF) | Day 1, measurements done immediately (within 1 hour) before and after the intervention
  Difference in change between real and sham group, in intracortical facilitation (ICF) measured with paired-pulse TMS-EMG.
  The ICF is the ratio between the amplitude of a motor-evoked potential from 2 TMS pulses delivered at 80% and 120% of the resting motor threshold at an interval of 10ms, and a control potential evoked by a single pulse at 120% of resting motor threshold.
Change across 1 intervention session in TMS-evoked recruitment curve at rest | Day 1, measurements done immediately (within 1 hour) before and after the intervention
  Difference in change between real and sham group, in characteristics of at-rest recruitment curve, measured with single-pulse TMS-EMG.
  A recruitment curve is the characteristic input/output relationship between stimulation-intensity of the TMS-pulse and the amplitude of the motor-evoked potential.
Change across 1 intervention session in TMS-evoked recruitment curve at slight tonic contraction | Day 1, measurements done immediately (within 1 hour) before and after the intervention
  Difference in change between real and sham group, in characteristics of recruitment curve at slight tonic contraction, measured with single-pulse TMS-EMG.
  A recruitment curve is the characteristic input/output relationship between stimulation-intensity of the TMS-pulse and the amplitude of the motor-evoked potential.
Change across 1 intervention session in TMS-induced cortical silent period | Day 1, measurements done immediately (within 1 hour) before and after the intervention
  Difference in change between real and sham group, in the duration of the TMS-induced cortical silent period of the EMG-trace, measured in the hand contralateral to the stimulation site.
Change across 1 intervention session in TMS-induced ipsilateral silent period | Day 1, measurements done immediately (within 1 hour) before and after the intervention
  Difference in change between real and sham group, in the duration of the TMS-induced ipsilateral silent period of the EMG-trace. Ipsilateral meaning the reduction in EMG-activity in the measured muscle on the same side of the participant as the stimulation site.
Change from baseline in participant-reported fatigue severity, measured by a fatigue diary | Week after intervention, compared to week before intervention
  Difference in change in day-to-day fatigue measured using a diary of fatigue scores, filled out by each subject at home in the week before/after the intervention week.
  The diary consists of a VAS-fatigue scale, as well as a rating for distribution between physical and cognitive fatigue. It is adapted from other sources.
Change from baseline in participant-reported sleep quality, measured by a fatigue diary | Week after intervention, compared to week before intervention
  Difference in change in sleep quality according to fatigue diary. As part of the fatigue diary, each patient will be asked each morning for the approximate hours of sleep and the quality of their sleep.
Change from baseline in daily activity levels, measured by a wrist-borne accelerometer | Week after intervention, compared to week before intervention
  Difference in change in stepcount based on data from wearable accelerometer, worn by each subject at home in the week before/after the intervention week.
Change from baseline in Sleep quality, measured by a wrist-borne accelerometer | Week after intervention, compared to week before intervention
  Difference in change in sleep efficiency, as assessed based on data from wearable accelerometer, worn by each subject at home in the week before/after the intervention week.
Effective dose at target brain region, calculated through E-field simulation | Intervention Days 1-5
  Exploratory. Simulated effective electric field dose at the targeted brain region (PMd), based on the individual pulse stimulation locations and an individual head-model based on subject-specific MR images. Simulated using SimNIBS.
  Exploratory analysis of whether actual stimulation intensity drives a potential positive treatment effect.

CONTACTS AND LOCATIONS:
Overall Officials: Hartwig R Siebner, MD, DMSc, Principal Investigator — Danish Research Centre for Magnetic Resonance, Copenhagen University Hospital Hvidovre & University of Copenhagen
Locations (1):
- Danish Research Centre for Magnetic Resonance, Hvidovre, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No
In accordance with Danish data protection legislation, it is currently not allowed to publish individual participant data.
  Data that underlie published results related to the primary and secondary outcome measures will, following anonymization, be made available upon reasonable request. However, data will be grouped in appropriate age categories with minimum 5 participants in each group.